CLINICAL TRIAL: NCT05320315
Title: Protective Effect Assessment Foto Ultra Isdin Solar Allergy Fusion Fluid (Isdin, s.a.) on the Ultraviolet A Induced Polymorphic Light Eruption
Brief Title: Protective Effect Assessment of Foto Ultra Isdin Solar Allergy Fusion Fluid on the UVA Induced PLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Pharmacologie Clinique Applique a la Dermatologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISD-FT-355-01-2020
Record Dates: First submitted 2021-09-17; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Polymorphic Light Eruption

STUDY DESIGN:
Intervention Model Description: Monocentric, single-blind, randomized, controlled, study with intra-individual comparisons
Masking Description: The study was Investigator evaluator blinded. The products were dispensed according to the randomization list by a responsible designated person other than the Investigator evaluator and/or evaluators. The randomization list was masked to the Investigator evaluator during the whole study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACTIVE and UNTREATED (Other): This was an intraindividual comparison study. Active (DM sunscreen) treated zone and Untreated zone are compared
  Interventions: Device: Foto Ultra ISDIN® Solar Allergy Fusion Fluid

INTERVENTIONS:
Device: Foto Ultra ISDIN® Solar Allergy Fusion Fluid — The tested MD is a very high protection sunscreen

SUMMARY:
The primary objective of this Clinical Investigation was to assess the protective efficacy of a medical device (FOTO ULTRA ISDIN® SOLAR ALLERGY FUSION FLUID) against the polymorphic light eruption induced by the UVA.

The secondary objective of this Clinical Investigation was to assess the local safety and the overall tolerability of the test MD on the basis of AE/SAE reporting.

DETAILED DESCRIPTION:
This was a PMCF investigation for a MD CE marked and used in its intended purpose with additional procedure non-invasive or non-burdensome.

This was a monocentric, single-blind, randomized, and controlled study performed with intra-individual comparisons. It is a type 2 Interventional study with minimal risks and constraints.

At least Fifteen (15) subjects with a known history of typical PLE on the chest after intense sun exposure were included in the study. The subjects were recruited via the CPCAD Subject Database or from those who spontaneously come to the CPCAD.

At Day 1, the tested MD was applied (2mg/cm²) on on side (10x15cm area) of the chest of each subject. The other side was not treated. Then, 15 minutes after application, both sides were irradiated with 40L/cm² of UVA. Same procedure was used from Day 2 to Day 5 with inceased UVA dose at Day 3 and Day 4 (50J/cm²) and Day 5 (60J/cm²).

UVA exposures have to be stopped once a PLE reaction was induced. Assessments (clinical, colorimetrical and photographs) were performed each day. Last assessments were perfomed at Day 8.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes aged >18 years with a known history of typical PLE on the chest after intense sun exposure and a last PLE outbreak since at least eight months,
2. Subject with Phototype I to IV according to the Fitzpatrick classification (1988) (14),
3. Subject in good health having normal results for the physical examination and medical antecedents compatible with the study requirements,
4. subject of non-childbearing potential (tubal ligation, hysterectomy, bilateral ovariectomy), or, subject of childbearing potential who has been, in the opinion of the Investigator, using an approved method of birth control (e.g. oral contraception pill or patch, intra-uterine devices, contraceptive implants or vaginal rings, condoms, bilateral tubal ligation) for at least 1 month prior to first visit. Subject must agree to continue adequate contraception during the entire study period and for 1 month after the end of the study,
5. Subject who, in the Investigator's opinion, will comply with the requirements of the protocol (e.g., follow protocol instructions, maintain regular contact to allow evaluation during the study),
6. Subject agreeing to avoid exposure to UV radiation (tanning beds, phototherapy, and sunlight) on the whole body for at least six months before the screening visit and for the whole duration of the study,
7. Subject agreeing to not apply cosmetic, medical or aesthetic treatments out of the study protocol on the chest during the whole study duration,
8. Healthy subject registered with Social Security in accordance with French law on interventional research. (Law 2004-806 and its implementing decree n°2006-477 of 26 April 2006).

Exclusion Criteria:

1. Female subject who is pregnant, parturient or breast feeding,
2. Subject of childbearing potential having a positive urinary pregnancy test at Day 1,
3. Subject has a PLE outbreak in the past eight months,
4. Subject has a medical condition or is taking medication that could put him or her at undue risk,
5. Subject has a pathology that is unstable or risks interfering with the study,
6. Subject is currently receiving treatment that may interfere with interpretation of the study results,
7. Subject has known or suspected allergies or sensitivities to any of the components of the study product,
8. Subjects with an underlying pathology, or with a surgical, physical or medical status which, according to the investigator, could interfere with the interpretation of the study results such as:

   1. Dermatological active pathologies (e.g. acne, psoriasis, eczema, urticaria...) in particular on the tested area (the chest) or suspicion/antecedents of allergies to cosmetics,
   2. All systemic or local uncontrolled pathologies,
   3. S kin anomalies (scars, excessive hair, tattooing…) on the chest,
9. Subjects having been exposed to ultraviolet radiation (UV), natural (sun) or artificial (tanning salon), in the 6 months before the initial visit or who plans such an exposure during the study,
10. Subjects having taken a systemic treatment, able to induce an abnormal response to UV, for more than 5 days during the month preceding inclusion (steroids, non-steroidal anti-inflammatories such as aspirin, insulin, antihistamines, anti-hypertensives, antibiotics such as quinolones, tetracyclines, thiazides and fluoroquinolones, and all other photosensitising treatments) or all treatments capable of inducing an abnormal response to UV (vitamin A derivatives, psoralen, aminolevulinic acid derivatives…) or planning to take these treatments during the study,
11. Subjects having applied a local treatment on the chest for more than 2 days during the 2 weeks preceding inclusion (steroids, non-steroidal anti-inflammatories, antihistamines, antibiotics) and all other cosmetic products in the previous 24 hours,
12. Protected subject as defined in the Articles of the CSP: Article 1121-7: person deprived of liberty by a judicial or administrative decision, or subject to psychiatric care or person admitted to a health or social institution for purposes other than the research. Article 1121-8: adult person subject to a legal protection measure or unable to express his/her consent.
13. Subject unable to communicate or cooperate with the Investigator due to poor mental development, language problems or impaired cerebral function,
14. Subject currently participating in another clinical study related to pharmaceuticals or MDs or being in an exclusion period of another clinical study,
15. Subject who has received (or who will receive) more than 4500 euros as indemnity for participating in clinical studies within the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Cumulative number of subjects who don't develop a positive PLE reaction | Day 8
  Cumulative number of subjects who don't develop a positive PLE reaction (at Day 8)

SECONDARY OUTCOMES:
Cumulative number of subjects who don't develop a positive PLE reaction by day | from Day 1 to Day 8
  Cumulative number of subjects who don't develop a positive PLE reaction by day
PLE severity score | from Day 1 to Day 8
  Scale of severity of polymorphous light eruption, 0 (no PLE) to 3 (severe PLE)

OTHER OUTCOMES:
Colorimetry component a* | from Day 1 to Day 8
  component a* related to erythema

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD, Nice, Cpcad, France

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Duteil L, Queille-Roussel C, Aladren S, Bustos X, Trullas C, Granger C, Krutmann J, Passeron T. Prevention of Polymorphic Light Eruption Afforded by a Very High Broad-Spectrum Protection Sunscreen Containing Ectoin. Dermatol Ther (Heidelb). 2022 Jul;12(7):1603-1613. doi: 10.1007/s13555-022-00755-5. Epub 2022 Jun 18. PMID 35716331